CLINICAL TRIAL: NCT05121077
Title: A Prospective, Comparative Analysis of Moderate-continuous (MCT) and Interval Training (IT) in LVAD (Left Ventricular Assist Device) Patients With Terminal Heart Failure: Train the LVAD Trial
Brief Title: Interval Versus Continuous Training in LVAD Patients
Acronym: TrainLVAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Peter Lüdike, Prof., University Hospital, Essen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-10169-BO
Record Dates: First submitted 2021-10-23; First posted 2021-11-16 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Heart Failure
Keywords: Exercise capacity; VO2peak; Interval training
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either the MCT or IT training group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate continuous training (Experimental): Participants will continuously exercise at a workload between 50-60% of VO2peak on a bicycle ergometer.
  Interventions: Other: Training
- Interval training (Experimental): Participants will exercise at a varying workload between 50-60% of VO2peak during recovery and 80-90% of VO2peak during bouts of interval training on a bicycle ergometer.
  Interventions: Other: Training

INTERVENTIONS:
Other: Training — 2 types of training intervention will be applied in terminal heart failure patients supported with a left ventricular assist device.

SUMMARY:
Patients with a left ventricular assist device (LVAD) will be randomized to either a moderate continuous (MCT, 50-60% of VO2peak) or interval training (IT, 80-90% of VO2peak) group for 6 weeks with 3 sessions per week, lasting for 20 minutes. An additional 10 minutes of resistance training will be performed in each group. Improvement of VO2peak and quality of life (KCCQ score) between the groups will be assessed.

DETAILED DESCRIPTION:
In- and out-patients with left ventricular assist device (LVAD) will be recruited to participate. On consent to participate, patients will be randomized to either moderate continuous (MCT) or interval (IT) training. An initial cardiopulmonary exercise test (CPET) will be performed to assess exercise intensity levels using a ramp protocol. Baseline quality of life (KCCQ score), echocardiographic and LVAD parameters, lab works, including NTproBNP, a 6min walk distance (6 MWD) will be assessed. Patients will then receive 6 weeks of supervised training in our facility (3x/week, 30min each). Following these sessions CPET, lab works, KCCQ assessment, 6 MWD, and echocardiography will be performed to assess improvement of exercise capacity.

Patients in the MCT group will receive 20min of moderate, continuous bicycle training at an intensity of 50-60% of VO2peak, the IT group will increase exercise density by increasing the duration of intense bouts (80-90% of VO2peak) over the weeks. All groups will receive an additional 10 minutes of resistance training (total exercise time 30 minutes in both groups). Improvement of VO2peak and quality of life (KCCQ score) between the groups will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years
* clinically stable LVAD patients with terminal heart failure
* written informed consent
* the mental and physical ability to exercise

Exclusion Criteria:

* established contraindications for exercise testing
* systemic blood stream infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-09-18 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Improvement of peak oxygen uptake (VO2peak) in cardiopulmonary exercise testing (CPET) [ml/kg/min] | 6 weeks
  Improvement of VO2peak in CPET after a training period of 6 weeks. CPET will be performed before (t0) and after (t1) the training period. A significant improvement from t0 to t1 is considered to be an increase of at least 2,5ml/kg/min

SECONDARY OUTCOMES:
Improvement in quality of life assessed by the Kansas City Cardiomyopathy Questionnaire (KCCQ) | 6 weeks
  Improvement in quality of life assessed by the Kansas City Cardiomyopathy Questionnaire (KCCQ) score. Points range from 0 to 100 in each of four domains. The total score is the average of all domains, with higher values depicting better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lüdike, Prof., Principal Investigator — Westdeutsches Herz- und Gefäßzentrum Essen, Klinik für Kardiologie und Angiologie
Locations (1):
- Uniklinikum Essen, Essen, Germany

IPD SHARING:
Plan to Share IPD: No
Individual data can be made available by the principal investigator on reasonable request.